CLINICAL TRIAL: NCT04114773
Title: Restoring Life After Cardiac Arrest - a Pilot Study of a Comprehensive Rehabilitation Intervention Focused on Fatigue for Survivors of Cardiac Arrest
Brief Title: Rehabilitation for Survivors of Cardiac Arrest Focused on Fatigue
Acronym: SCARF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: REHPA The Danish Knowledge Center for Rehabilitation and Palliative Care (Unknown); University of Southern Denmark (Other); Odense Patient Data Explorative Network (Other); Center for Rehabilitation of brain injury, Copenhagen (Unknown)
Responsible Party: Principal Investigator, Vicky Joshi, Principal investigator, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20192000-66
Record Dates: First submitted 2019-09-18; First posted 2019-10-03 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Arrest With Successful Resuscitation
Keywords: Rehabilitation; Fatigue; Relatives
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCARF (Experimental): The participants will take part in a rehabilitation intervention focused on the physical, mental, and social consequences of cardiac arrest with an overarching theme of managing fatigue. This will consist of:
  * a 5-day residential rehabilitation stay
  * followed by a 12 week home-based programme including one telephone call by a member of the clinical rehabilitation team,
  * after the 12 week home intervention there will be a further 2-day rehabilitation stay.
  Interventions: Other: SCARF (Survivors of Cardiac Arrest Rehabilitation focused on Fatigue)

INTERVENTIONS:
Other: SCARF (Survivors of Cardiac Arrest Rehabilitation focused on Fatigue) — The intervention will be delivered by a multidisciplinary team. There will be individual testing and feedback on physical capacity and cognitive ability. Group sessions will include education on the consequences of cardiac arrest, promotion of techniques to ameliorate these consequences, for example, increasing physical activity or energy conservation. Additional sessions will cover psychological reactions; family life; work life; intimacy; and existential considerations.
  Participants will have a course information book with a physical activity training diary and problem-solving therapy worksheets to use at home for 12-weeks. They will receive one phone call from the clinical team during this period. The 2-day return stay will revisit the subjects from the first 5-day stay.
  Participating survivors who have a relative that wishes to attend will be included in all the group sessions and individual feedback but will not take part in the physical capacity or cognitive ability tests.

SUMMARY:
More people are surviving a cardiac arrest due to improvements in bystander resuscitation and acute hospital care. However, many survivors of cardiac arrest are left with physical, mental and social problems impacting negatively on their quality of life. At present there are no specialist interventions for survivors of cardiac arrest in Denmark and very few have been evaluated internationally. Rehabilitation for people after cardiac events or brain injury have shown significant physical and mental well-being benefits, indicating the same may be true for survivors of cardiac arrest.

This pilot study will test the feasibility and acceptability of a residential rehabilitation intervention focused on fatigue, and the physical, mental and social consequences of cardiac arrest. In addition, the pilot study will discover if the intervention has any effect on self-report measures, including fatigue, mental well-being and activity of the survivors of cardiac arrest who participate, and on the mental well-being of relatives of these survivors.

DETAILED DESCRIPTION:
The number of people surviving a cardiac arrest is increasing every year due to advances in pre-hospital and acute medical care. In Denmark, one year survival after out-of-hospital cardiac arrest improved from 4-13% between 2001 and 2014; this amounts to at least 500 new survivors every year. But after the acute phase ends, many survivors of cardiac arrest (SCA) suffer an uncertain future. Most SCA will have a new or ongoing cardiac condition. They may suffer from mental trauma due to surviving a near death experience. Further, reduced oxygen levels to the brain during a cardiac arrest, can cause brain injury in up to 50% of SCA. This combination of cardiac, traumatic and neurological factors causes survivors to suffer from a wide range of physical, psychological and cognitive problems impacting negatively on their quality of life. Relatives of SCA have also been found to suffer from emotional problems due to becoming a carer for their loved one.

Normally in Denmark, a patient population with such a heavy burden, like SCA and their relatives would receive help to restore them to daily life but at present there are no specialist rehabilitation interventions provided for SCA in Denmark.

Research involving rehabilitation interventions for people after brain injury or cardiac events has shown significant physical, psychological and quality of life benefits, indicating the same may be true for SCA. The European Resuscitation Council and other international experts recommend all SCA receive rehabilitation tailored to their needs but very few research studies exist on which to base the design of these rehabilitation interventions.

The Medical Research Council (MRC) in the United Kingdom state that in clinical research there is too strong a focus on the main evaluation of an intervention. This means inadequate development and piloting work, leading to weaker interventions that are less likely to be implemented. Before performing large-scale testing of an intervention, the MRC advocates a systematic development phase that tests the feasibility of the new intervention.

Though examination of current literature and workshops with researchers, clinicians, survivors of cardiac arrest and their relatives a new comprehensive rehabilitation intervention has been developed.

The objectives of this study are to, firstly, test the feasibility and acceptability of the intervention. Secondly, to determine the effect of the intervention on patient reported outcomes covering fatigue, physical activity, psychological well-being and quality of life. In addition, the effect of the intervention on the mental well-being of any relatives who take part in the intervention.

Recruitment will take place via publicity through REHPA, the five cardiac centers in Denmark and via the Danish Heart Foundation. Potential participants will apply via an application form and be screened by the research team for eligibility.

ELIGIBILITY:
Inclusion Criteria:

* At least 3-months post-cardiac arrest
* Self-identified need for rehabilitation as measured by a score of 3 or above on the Dallund scale, a linear analog self-assessment scale, where participants indicate how close they are to living the life they desire after their cardiac arrest, indicating rehabilitation needs. The scale is rated between 0 (goal reached) and 10 (infinitely far from).
* Self-reliant with personal care and medication

Exclusion Criteria:

* Medical needs requiring in-patient medical treatment
* No permanent residence in Denmark
* Not able to speak and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate for participants | Time frame: From month 4 to month 1 before intervention start date
  Recruitment rate for participants (survivors and relatives), number of participants recruited per week.
Participant satisfaction assessed by a likert scale | At eleven weeks months
  Participant (survivors and relatives) satisfaction with intervention as assessed by a 5-point likert scale for each component of the intervention.
  In addition, qualitative interviews with participants (survivors and relatives)
Completion of study outcome measures | Baseline, eleven weeks and 6 months
  Percentage of participants (survivors and relatives) who complete each outcome measure
Adherence to intervention by participants | At eleven weeks
  Percentage of participants (survivors and relatives) who achieve minimum adherence levels, that is attendance at both the 5-day rehabilitation stay and 2-day follow-up rehabilitation stay.

SECONDARY OUTCOMES:
Efficacy of improving fatigue as measured by the change from baseline in the Modified Fatigue Impact Scale | Baseline, at eleven weeks, 6 months
  The Modified Fatigue Impact Scale assesses how fatigue impacts functional activities, the self-report questionnaire has 21 items in three sub-scales (physical, cognitive and psychosocial). Scores are summed to give a total. Total scores range from 0-84. The ranges of scores for each sub-scale are as follows: physical, 0 to 36; cognitive, 0 to 40; and psychosocial, 0 to 8. Higher scores indicate a greater impact of fatigue.
Efficacy of improving fatigue as measured by the change from baseline in the Multidimensional Fatigue Inventory | Baseline, at eleven weeks, 6 months
  The Multidimensional Fatigue Inventory measures fatigue severity, it covers five dimensions; general fatigue, physical fatigue, reduced activity, reduced motivation and mental fatigue. Higher scores indicate a higher level of fatigue, with 4 being no fatigue and 20 the worst imaginable fatigue
Efficacy of improving physical activity as measured by the change from baseline in the International Physical Activity Questionnaire Short | Baseline, at eleven weeks, 6 months
  The International Physical Activity Questionnaire Short is a self-report questionnaire that has 7 items providing information on time spent walking, in vigorous- and moderate- intensity activity. Total time spent performing activities is summed and results reported in categories low, medium and high physical activity levels.
Efficacy of improving activity and participant as measured by the change from baseline in the World Health Organisation Disability Assessment Schedule 2.0 | Baseline, at eleven weeks, 6 months
  The World Health Organisation Disability Assessment Schedule 2.0 is a self-report questionnaire that assesses disability and functioning in the prior month. It assesses six different adult life tasks: 1) Understanding and communication; 2) Self-care; 3) Mobility (getting around); 4) Interpersonal relationships (getting along with others); 5) Work and household roles (life activities); and 6) Community and civic roles (participation). There are 36 items scored from 0- no difficulty to 4- extreme difficulty or cannot do. Total scores range from 0 to 144 with a higher score indicating greater difficulty with activity and participation. Completed by survivors only.
Percentage of survivor participants who identified and solved the set minimum number of problems in the problem-solving therapy component of the intervention | At end of 2-day follow-up intervention phase, an average of 12 weeks.
  Minimum number of problems to be generated and solved during the intervention is two. A problem will be deemed identified and solved if each of the 7 stages in the written problem-solving therapy has been completed and the participant marks the problem as solved.
Percentage change in survivors '6 minutes walk test' from baseline to follow up (survivors) | Baseline and at follow-up after 11 weeks
  '6 minutes walk test' will be performed at baseline and follow-up. Measurements will be performed by trained health professionals and standardised protocols will be followed. The change in percent will be calculated for each individual survivor participant.
Percentage change in hand grip strength from baseline to follow up (survivors) | Baseline and at follow-up after 11 weeks
  Hand grip strength will be measured with a calibrated hand dynamometer at baseline and at follow up. Measurements will be performed by trained health professionals and standardised protocols will be followed. Three measurements will be performed for each participant and the mean will be calculated. The change in percent will be calculated for each individual participant.
Percentage change in '30 seconds sit-to-stand-test' from baseline to follow up (survivors) | Baseline and at follow-up after 11 weeks
  '6 minutes walk test' will be performed at baseline and follow-up. Measurements will be performed by trained health professionals and standardised protocols will be followed. The change in percent will be calculated for each individual participant.
Efficacy of improving anxiety and depression as measured by the change from baseline in the Hospital Anxiety and Depression Scale. To be completed by survivors and relatives. | Baseline, at eleven weeks, 6 months
  Description: The Hospital Anxiety and Depression Scale consists of a seven-item subscale for anxiety (HADS-A) and a seven-item subscale for depression (HADS-D), and is used to assess symptoms of anxiety and depression.. Each item has a four choice response with scores ranging from 0 for no symptoms to 3 for the maximum number of symptoms. The scores on each subscale range from 0 to 21.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Dorthe Zwisler, Professor, PhD, Study Director — REHPA The Danish Knowledge Center for Rehabilitation and Palliative Care
Locations (1):
- REHPA The Danish Knowledge Center for Rehabilitation and Palliative Care, Nyborg, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No